CLINICAL TRIAL: NCT06710691
Title: A Randomized Factorial Feasibility Study of High-Resistance Circuit Training and Strength Training Intervention in Untrained Adolescents: A Mixed Methods Approach
Brief Title: Feasibility Study of Resistance Training Intervention in Untrained Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Mitch Wyatt, PhD Student, University of Utah
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: IRB_00166762
Record Dates: First submitted 2024-11-20; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Feasibility Studies
Keywords: High-Resistance Circuit Training; Strength Training; Resistance Training; Feasibility; Mixed-Methods; Before-School; After-School

STUDY DESIGN:
Intervention Model Description: The study also used an explanatory sequential design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Before-school high-resistance circuit training group (Experimental): Participants conducted circuit-based training before school at submaximal intensities (6, 7 and 8 RPE) with limited rest between exercises.
  Interventions: Other: Physical activity intervention using high-resistance circuit training.
- Before-school strength training group (Active Comparator): Participants conducted strength training before school at submaximal intensities (6, 7 and 8 RPE) with 1 min rest between exercises.
  Interventions: Other: Physical activity intervention using traditional strength training protocols
- After-school high-resistance circuit training group (Experimental): Participants conducted circuit-based training after school at submaximal intensities (6, 7 and 8 RPE) with limited rest between exercises.
  Interventions: Other: Physical activity intervention using high-resistance circuit training.
- After-school strength training group (Active Comparator): Participants conducted strength training after school at submaximal intensities (6, 7 and 8 RPE) with 1 min rest between exercises.
  Interventions: Other: Physical activity intervention using traditional strength training protocols

INTERVENTIONS:
Other: Physical activity intervention using traditional strength training protocols — Strength training participants performed the 6 reps of the first exercise at the prescribed RPE and then rested for 1 minute. Participants then completed another set of their first exercise with the required rest until the prescribed sets were completed. Participants performed the second and third exercises in the same fashion. Once the first block was completed, participants rested 5 min, then completed the second block. Six exercises were completed.
  Other Names: ST
  Arms: After-school strength training group; Before-school strength training group
Other: Physical activity intervention using high-resistance circuit training. — An adapted version of Alcaraz's high-resistance circuit training (HRC) was utilized in the intervention. Exercises and intensities used by strength training was the same for HRC except HRC participants performed the first three exercises as a circuit with 35 seconds rest between exercises, then completed the second block of exercises in the same fashion.
  Arms: After-school high-resistance circuit training group; Before-school high-resistance circuit training group

SUMMARY:
Adolescents may have limited time to engage in physical activity during the school day prompting investigations of before and after-school times along with time efficient programming. High-resistance circuit training has been used as a time effective protocol, however adolescents have yet to be studied. The primary aim was to assess feasibility (recruitment, sample size, consent rate, retention rate, fidelity, attendance, adverse events, and participant experience) of a high-resistance circuit training or strength training intervention, conducted before or after-school. The second aim was to explore changes in body composition, strength, and aerobic fitness.

Researchers compared feasibility outcomes as well as participant experience between time frames and treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Untrained
* Male and female
* Student at site
* Available to workout before or after-school

Exclusion Criteria:

* Recent injuries or medical conditions that may influence high-intensity performance
* Currently enrolled in another training program including resistance, cardiovascular, or sports-based program
* Uninsured participants
* Drastically altering diet
* Use of performance-enhancing substances (i.e., creatine, pre-workout, post-workout supplements).

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Recruitment process | Three weeks.
  The recruitment process refers to the protocols used to find, select, and enroll participants into a study. The recruitment process for this study was represented by reporting the total number of unique QR code scans from posted flyers and tabling events, the number of completed interest forms, the number of eligible participants and the number of consented participants. A recruitment period of 3 weeks was given for the before and after-school trials.
Sample Size | From enrollment through 4 weeks of treatment.
  Sample size was used as another key feasibility marker and refers to the total number of individuals used in the intervention.
Consent Rate | From a 3 week recruitment period to enrollment.
  Consent rate is often referred to as the percentage of participants enrolled divided by the number of eligible participants. For this study, consent rate was calculated by taking the total number of participants that consented and were randomized divided by the number of eligible students.
Retention Rate | From enrollment through 4 weeks of treatment.
  Retention rate is defined as the percentage of the total number of randomized participants assessed for primary outcomes and used in the primary outcome analysis. For the purpose of this study, researchers were interested in retention for both primary and secondary outcomes meaning researchers tracked retention from pre-intervention fitness testing, through treatments, and post-intervention fitness testing sessions. The follow up interview was not included in calculating the retention rate. Only participants that withdrew from the study or were not included in the primary and secondary outcome analysis influenced the retention rate. Thus, retention was calculated as the percentage of participants that completed pre and post-intervention fitness assessments and intervention treatment divided by the number of participants randomized into treatment groups.
Fidelity | From enrollment through 4 weeks of treatment.
  For this study, fidelity was assessed at the instructor and participant level. Instructor fidelity was measured as a percentage by totaling the provided sessions divided by the total number of planned sessions. An acceptable percentage was set at 80% due to conflicts with events such as holiday breaks or parent teacher conferences. To assess participant fidelity, the primary researcher and participants recorded session durations, completed sets and intensity along with activity and diet audits at weeks 2, and 4 of the intervention. The activity and diet audit included a modified Copper Institute Fitnessgram and Activitygram questionnaire.
Average Attendance | From enrollment through 4 weeks of treatment.
  Participant attendance was observed by the researcher and measured as attended sessions divided by total sessions offered.
Adverse Events | From enrollment through 4 weeks of treatment.
  Adverse events were recorded during the intervention by the participants on workout documents and by observations from the primary researcher.
Participant Experience | From enrollment through 4 weeks of treatment in addition to a 1 month follow up interview.
  Participant experience was assessed by utilizing the validated short form 4 item Physical Activity Enjoyment Scale (PACES-S) survey for adolescents [48]. Participants answered 4 items including: "I enjoyed it; I find it pleasurable; It is very pleasant; and It feels good" by responding with the five-point Likert scale ranging from 1= "strongly disagree" to 5 = "strongly agree". To further investigators' depth of understanding, participant experience was also assessed by a follow up interview concluding the intervention.

SECONDARY OUTCOMES:
Body Mass Index | Through study completion, an average of 4 weeks
  In a separate private room, one participant at a time weighed themselves on a certified scale. Participants used the handheld Omron model HBF-306 to enter their weight, age, sex and activity level. Resulting body mass index (kg/m^2) was recorded.
Body Fat Percentage | Through study completion, an average of 4 weeks
  In a separate private room, one participant at a time weighed themselves on a certified scale. Participants used the handheld Omron model HBF-306 to enter their weight, age, sex and activity level. Resulting body fat percentage data was recorded.
Isometric lower body pull | Through study completion, an average of 4 weeks
  Isometric lower body pull. Using the Baseline 12-0400 Back-Leg-Chest dynamometer participants stood up-right and feet hip width apart on the dynamometer platform with the chain adjusted so the handle was at the intra-articular space of the knee joint. Participants were instructed to grip the handle evenly at the center then produce a maximal 5 sec pull keeping the back from bending and arms straight. Participants were allowed to rest 30 sec between attempts. Participants had one practice attempt for familiarization purposes and then the best score of the three following attempts were recorded.
90° push-up | Through study completion, an average of 4 weeks
  Participants were paired; participant 1 performed the test while participant 2 recorded the number of push-ups. Participants performed the assessment in accordance with the Cooper Institute's procedures. Participant 1 assumed a prone plank position with hands slightly outside of shoulders, fingers stretched out and legs straight with a slight gap. While performing push-ups, the participants' back maintained a straight line from head to ankles. Participants started by lowering their body until the upper arms became parallel to the ground. The participant then extended their arms straight pushing their body up. This movement was performed every three seconds by metronome and repeated until failure. Participants were allowed one form correction and two form corrections resulted in test termination. Form corrections included participants stopping to rest, a failure to maintain a straight back, achieving proper depth or fully extending the arms.
Modified Pull-up | Through study completion, an average of 4 weeks
  Participants performed the modified pull-up test in accordance with Cooper Institute's procedure. Participants placed a barbell in a squat rack so that the barbell was one to two inches away from participant's reach while supine on the ground. A band was then placed seven to eight inches below the barbell. Participants started the assessment by overhand gripping the barbell and creating a straight line from head to heels so that only the heels were in ground contact. Participants then pulled their body toward the barbell until the chin was above the band. This movement was performed every three seconds by metronome and repeated until failure. Participants were allowed one form of correction and two form corrections would result in test termination. Form corrections included participants stopping to rest, failure to maintain a straight line, achieve proper depth and fully extending the arms.
Aerobic Fitness | Through study completion, an average of 4 weeks
  To assess cardiovascular fitness, the Progressive Aerobic Cardiovascular Endurance Run (PACER) assessment was used. Prior to the start of assessment, the primary investigator measured and marked a designated 20-meter distance in the gymnasium for testing. Participants were briefed on the assessment guidelines and participated in one practice opportunity prior to the official assessment. Once familiarized, participants ran the 20-meter distance in accordance to PACER cadences from the Cooper Institute for as long as possible. The test was terminated when the participant voluntarily stopped due to fatigue or when two laps were missed. The primary researcher recorded total number of successful levels. Once completed, the primary researcher computed predicted peak VO2 by using VO2peak = 0.353(Laps) - 1.121(Age) + 45.619.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Brusseau Jr., Study Chair — University of Utah
Locations (1):
- Murray High School, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No
In the consent process, participants and guardians were informed that their data will not be used in future studies.

DOCUMENTS (7):
  • Study Protocol and Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT06710691/Prot_SAP_000.pdf
  • Informed Consent Form: Before-School Informed Consent Form (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT06710691/ICF_001.pdf
  • Informed Consent Form: Before-School Assent Form (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT06710691/ICF_002.pdf
  • Informed Consent Form: Before-School Parental Permission Form (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT06710691/ICF_003.pdf
  • Informed Consent Form: After-School Consent Form (2023-10-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT06710691/ICF_004.pdf
  • Informed Consent Form: After-School Assent Form (2023-10-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT06710691/ICF_005.pdf
  • Informed Consent Form: After-School Parental Permission Form (2023-10-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT06710691/ICF_006.pdf